CLINICAL TRIAL: NCT04009044
Title: A Phase II Study of the Determinants of Transdermal Drug Delivery to the Normal and the Radiated Breast
Brief Title: Topical Afimoxifene in Treating Patients With Breast Cancer Who Have Undergone Radiation Therapy on One Breast
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 18B05; NCI-2019-03771 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NU 18B05 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Cancer Survivor; Ductal Breast Carcinoma In Situ; Invasive Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — afimoxifene; 4,17 beta-dihydroxy-4-androstene-3-one; Biopsy, Needle; Biopsy, Large-Core Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (afimoxifene) (Experimental): Patients apply afimoxifene gel topically QD to both breasts for 3 to 5 weeks and then undergo core needle biopsies of both breasts.
  Interventions: Drug: Afimoxifene; Procedure: Core Biopsy; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Afimoxifene — Apply topically
  Other Names: 4-Hydroxy-Tamoxifen; 4-hydroxytamoxifen; 4-OHT
Procedure: Core Biopsy — Undergo core needle biopsy
  Other Names: core needle biopsy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well topical afimoxifene works in treating patients with breast cancer who have undergone radiation therapy on one breast. Topical afimoxifene is a quick-drying medicated gel that may block the growth of breast cancer cells when applied to the breast skin. The purpose of this research is to determine what effect, if any, differences in skin type between women have on the delivery of topical afimoxifene to the breast tissue, and whether radiation affects the delivery of topical afimoxifene to breast tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the skin features that drive inter-individual variation in dermal drug permeation between individuals.

SECONDARY OBJECTIVES:

I. To relate breast tissue drug concentration to skin histology, skin vascularity, skin transporter proteins, and skin features measured using confocal reflectance microscopy.

II. To assess the feasibility of transdermal drug delivery to the radiated breast.

OUTLINE:

Patients apply afimoxifene gel topically once daily (QD) to both breasts for 4 weeks and then undergo core needle biopsies of both breasts.

Patients receive follow up phone call 21-35 days after biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received prior unilateral breast radiotherapy (RT) for ductal breast carcinoma in situ (DCIS) or invasive cancer (>= 12 weeks after the end of RT), and have an intact unradiated (non-RT) breast.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%).
* A prior history of malignancy is allowed, as long as the patient is considered to have ?no evaluable disease? and cancer treatment has been completed.
* Females of child-bearing potential (FOCBP) and male partners of female participants must agree to use TWO effective forms of birth control (abstinence is not an allowed method) prior to study entry and for the duration of study participation, and for two months following the last dose of study medications. Effective birth control methods are: copper IUD (intrauterine device), diaphragm/cervical cap/shield, spermicide, contraceptive sponge, condoms. Should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months).
* FOCBP must have a negative urine pregnancy test within 7 days prior to registration on study.
* Willingness to avoid exposing breast skin to natural or artificial sunlight (i.e. tanning beds) for the duration of the study drug use.
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.

Exclusion Criteria:

* Patients receiving any other investigational agents within 30 days of registration are not eligible.
* Patients currently using oral selective estrogen receptor modulators (SERMS) (tamoxifen, raloxifene, bazedoxifene) are not eligible.

  * Note: Prior or current endocrine therapy other than SERMs are allowed.
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition afimoxifene (4-OHT) are not eligible.
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Hypertension that is not controlled on medication
  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient?s safety or study endpoints.
* Female patients who are pregnant or nursing are not eligible.
* Patients with prior bilateral breast cancer radiotherapy or radiotherapy for lymphoma will be excluded.
* Patients with skin lesions on the breast that disrupt the stratum corneum (e.g. eczema, ulceration) are not eligible.
* Patients with a history of endometrial neoplasia are not eligible.
* Patients with a history of thromboembolic disease are not eligible.

  * Note: history of varicose veins and superficial phlebitis is allowed.
* Patients who are undergoing active treatment for any malignancy will be excluded.
* Male patients are excluded from this study since there are no data regarding skin penetration of 4-OHT though male chest wall skin (which is thicker and hairier than female chest wall skin).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Determinants of inter-individual variation in afimoxifene drug concentrations in unradiated breast tissue related to skin histology, blood and lymph vessel density | Up to 35 days post-treatment
  Univariate analyses will relate each characteristic to tissue drug concentration using either correlation analysis for continuous characteristics or a t-test, analysis of variance or rank sum test for categorical characteristics. Multiple linear regression modelling will be used to select those characteristics that provide the strongest independent contribution to the model.
Determinants of inter-individual variation in afimoxifene drug concentrations in unradiated breast tissue related to the expression of xenobiotic transporters and enzymes | Up to 35 days post-treatment
  Univariate analyses will relate each characteristic to tissue drug concentration using either correlation analysis for continuous characteristics or a t-test, analysis of variance or rank sum test for categorical characteristics. Multiple linear regression modelling will be used to select those characteristics that provide the strongest independent contribution to the model.
Determinants of inter-individual variation in afimoxifene drug concentrations in unradiated breast tissue related to skin features | Up to 35 days pot-treatment
  Will be measured with confocal reflectance microscopy. Univariate analyses will relate each characteristic to tissue drug concentration using either correlation analysis for continuous characteristics or a t-test, analysis of variance or rank sum test for categorical characteristics. Multiple linear regression modelling will be used to select those characteristics that provide the strongest independent contribution to the model. A similar analysis will be conducted using the skin characteristics from the confocal reflectance microscopy.

SECONDARY OUTCOMES:
Effect of breast radiotherapy on drug concentrations resulting from transdermal delivery of afimoxifene (4-OHT) | Up to 35 days post-treatment
  Tissue drug concentrations will be compared between radiated and non-radiated breasts using a mixed linear model, with breast radiation status as a fixed effect of interest and person as a random effect. Analyses will also be done to compare the skin data (histology, immunohistochemistry [IHC], protein expression, CRS) between radiated and non-radiated breasts. While most characteristics will be continuous, other metrics will be analyzed by using different link functions in similarly constructed generalized linear model.
Differences between radiated and non-radiated skin and breast tissue that contribute to differences in permeation | Up to 35 days post-treatment
  Tissue drug concentrations will be compared between radiated and non-radiated breasts using a mixed linear model, with breast radiation status as a fixed effect of interest and person as a random effect. Analyses will also be done to compare the skin data (histology, IHC, protein expression, CRS) between radiated and non-radiated breasts. While most characteristics will be continuous, other metrics will be analyzed by using different link functions in similarly constructed generalized linear model.

CONTACTS AND LOCATIONS:
Overall Officials: Seema A Khan, M.D., Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois

REFERENCES:
- [Derived] Lee O, Pilewskie M, Karlan S, Tull MB, Benante K, Xu Y, Blanco L, Helenowski I, Kocherginsky M, Yadav S, Hosseini O, Hansen N, Bethke K, Muzzio M, Troester MA, Dimond E, Perloff M, Heckman-Stoddard B, Khan SA. Local Transdermal Delivery of Telapristone Acetate Through Breast Skin, Compared With Oral Treatment: A Randomized Double-Blind, Placebo-Controlled Phase II Trial. Clin Pharmacol Ther. 2021 Mar;109(3):728-738. doi: 10.1002/cpt.2041. Epub 2020 Oct 25. PMID 32996592